CLINICAL TRIAL: NCT06583967
Title: The Effect of Aerobic Exercise on an Elliptical Trainer Versus a Treadmill, on Gait and Walking Abilities, Expressed in Dynamic Stability, Balance and Walking Speed, in People With Multiple Sclerosis (MS)
Brief Title: The Effect of Aerobic Exercise on an Elliptical Trainer Versus a Treadmill, in People With Multiple Sclerosis
Acronym: MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Soroka University Medical Center (Other)
Responsible Party: Principal Investigator, Iuly Treger, M.D., PhD, MHA, Principal Investigator, Head of Rehabilitation Department, Soroka University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0104-23-SOR; 0104-23-SOR (Other: Soroka Medical Center, Ethics Committee)
Record Dates: First submitted 2024-08-27; First posted 2024-09-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2024-08

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Aerobic; Exercise; Elliptical trainer; Treadmill; 6 Minute Walk Test (6MWT); Timed Up & Go (TUG); Berg Balance Scale (BBS); 10 Meter Walk Test (10MWT); Informed Consent Form (ICF)
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity | interventions — Physical Conditioning, Human

STUDY DESIGN:
Intervention Model Description: The study will assess the effect of 12 weeks of aerobic exercise on an elliptical trainer (group 1) vs a treadmill (group 2), on gait and walking abilities, expressed in dynamic stability, balance and walking speed, in people with Multiple Sclerosis.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - Elliptical Trainer (Experimental): 15 MS subjects will be enrolled and assigned to group 1 and to be trained (Elliptical Trainer) twice a week for 12 weeks.
  Interventions: Other: Physical Training
- Group 2 - Treadmill (Experimental): 15 MS subjects will be enrolled and assigned to group 2 and to be trained (Treadmill) twice a week for 12 weeks.
  Interventions: Other: Physical Training

INTERVENTIONS:
Other: Physical Training — Group 1 - Elliptical Trainer Group 2 - Treadmill

SUMMARY:
The aim of this study is to examine the effects of aerobic exercise training using an elliptical trainer compared to a treadmill on gait and walking abilities, expressed in dynamic stability, balance, and walking speed, in people with Multiple Sclerosis with moderate severity.

DETAILED DESCRIPTION:
A total of 30 MS subjects to be enrolled in the study. Subjects to be assigned into one of two groups named: Group 1 - Elliptical Training and Group 2 - Treadmill Training. Effort capacity will measured by heart rate and RPE.

Outcome measures will be measured by using, 6 min. walking test (6MWT), Timed Up & Go (TUG), Berg Balance Scale (BBS) and 10 Meter Walk Test (10MWT) to be used to assess the quality of life at Baseline (T0), During study - 6 weeks from baseline (T1), End of training program - 12 weeks from baseline (T2) and 6 weeks post T2 (T3).

The exercise program to be applied for 12 weeks with 2 trainings per week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients signed Informed Consent Form
2. At least 6 months post MS diagnosis
3. 25-55 years old adults
4. EDSS 3.0-6.5
5. Standing stability - for at least 30 seconds
6. 6MWT - minimal distance to be measured as 210 meters
7. No physical routinely training e.g. walking, elliptical or cycling within 3 months prior screening visit.

Exclusion Criteria:

1. Active Heart Disease
2. Lungs and/or respiratory system diseases
3. Metabolic Disease
4. Any other medical condition(s) which might impact the patient's participant in the study, as per PI medical judgement
5. Major medical treatment change (as per PI medical judgement) up to 12 weeks prior ICF signature by the patient.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Quality of life outcomes | Baseline (screening), T1 (Week 6), T2 (Week 12), T3 (Follow-up, 6 weeks post T2)
  Quality of life to be assessed by using a Short-form 36 health status questionnaire (SF-36). SF-36 consists of 36 questions in total. Each participant will be asked to fill in the questionnaire alone and by reading it themselves.

SECONDARY OUTCOMES:
6 Minute Walk Test (6MWT) | Baseline (screening), T1 (Week 6), T2 (Week 12), T3 (Follow-up, 6 weeks post T2)
  Each subject will be asked to perform a 6 min walk and the max distance to be measured,
Timed Up & Go (TUG) | Baseline (screening), T1 (Week 6), T2 (Week 12), T3 (Follow-up, 6 weeks post T2)
  Patients wear their regular footwear and can use a walking aid, if needed. The patient stands up upon therapist's command: walks 3 meters, turns around, walks back to the chair and sits down. The time stops when the patient is seated
Berg Balance Scale (BBS) | Baseline (screening), T1 (Week 6), T2 (Week 12), T3 (Follow-up, 6 weeks post T2)
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks.
10 Meter Walk Test (10MWT) | Baseline (screening), T1 (Week 6), T2 (Week 12), T3 (Follow-up, 6 weeks post T2)
  The 10 Metre Walk Test is a performance measure used to assess walking or gait speed in meters per second over a short distance

CONTACTS AND LOCATIONS:
Overall Officials: Iuly Treger, MD, PhD, Principal Investigator — Soroka University Medical Center
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba, Israel
  - Israel ParaSport Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No
There isn't any plan to make IPD available to other researchers.